CLINICAL TRIAL: NCT03744663
Title: A Randomized Pilot Study of Long Acting Buprenorphine Injection Compared to Sublingual Buprenorphine/Naloxone Films
Brief Title: Long Acting Buprenorphine Injection Compared to Sublingual Buprenorphine/Naloxone Films
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding for uninsured subjects could not be realized and staffing after COVID hit was also a problem.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00054516
Record Dates: First submitted 2018-11-09; First posted 2018-11-16 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Opioid Use
Keywords: opioid; Opioid Agonist Treatment; buprenorphine; substance abuse; drug; abstinence
MeSH Terms: conditions — Substance-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination; Sublocade

STUDY DESIGN:
Intervention Model Description: Patients admitted to the WFBMC Medication-Assisted-Therapy (MAT) clinic with a diagnosis of moderate/severe Opioid-Use Disorders (OUD) who are more than 18 years old will be approached for enrollment in this study. Because of the nature of a pilot study, it's proposed a total of 30 patients, 15 in each group. Subjects will be started and titrated to optimal Suboxone® SL dose for 14 days. After the 14 day, the subject will be started on the treatment to which they are randomized, either Suboxone® SL or Sublocade®. Control group -Suboxone®SL: Patients assigned to this group will continue with their already established dose of Suboxone ®SL films for 24 weeks along with weekly therapy. Study drug-Sublocade® group: Patients assigned to this group will receive the study drug (subcutaneously) every 4 weeks for a total of 6 doses along with weekly therapy. At the end of the 24-weeks subjects will continue the medication of their choice within the constraints of their insurance provider.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Suboxone® SL (Active Comparator): Patients assigned to this group will continue with their already established dose of Suboxone ® SL films for 24 weeks along with weekly therapy.
  Interventions: Drug: Suboxone® SL
- Sublocade® (Experimental): Patients assigned to the Sublocade® group will receive the study drug (300 mg subcutaneously) every 4 weeks for a total of 6 doses along with weekly therapy.
  Interventions: Drug: Sublocade®

INTERVENTIONS:
Drug: Suboxone® SL — Subjects will be started and titrated to optimal Suboxone® SL dose for 14 days. After the 14 day induction phase, the subject will be started on the treatment to which they were randomized to two groups one of which will be Suboxone® SL.
  Other Names: Suboxone® SL films; buprenorphine naloxone
  Arms: Suboxone® SL
Drug: Sublocade® — Subjects will be started and titrated to optimal Suboxone® SL dose for 14 days. After the 14 day induction phase, the subject will be started on the treatment to which they were randomized, either Suboxone® SL or Sublocade®. Subjects with significant opioid craving (> 20 mm on the Opioid Craving Visual Analog Scale) or withdrawal (a score of > 12 on the Clinical Opiate Withdrawal Scale) after 14 days of treatment will be started on Sublocade® only at the consensus of the research team. Otherwise they will undergo an additional 7 day titration period. Study drug with Sublocade® group: Patients assigned to this group will receive the study drug (300 mg subcutaneously) every 4 weeks for a total of 6 doses along with weekly therapy. The location and specifications of its application will follow the recommendations by the FDA previously published.
  Other Names: buprenorphine extended-release
  Arms: Sublocade®

SUMMARY:
While substance use disorders have been found to have relapse rates on part with other chronic illnesses such as hypertension and asthma long term abstinence remains elusive for many. The FDA has recently approve a long acting subcutaneous injectable formulation of buprenorphine. This study aims to determine the feasibility of enrolling and randomizing patients seeking treatment at an outpatient substance abuse clinic to buprenorphine/naloxone films which dissolve under the tongue vs. long acting buprenorphine injection with all other treatment aspects held constant. The study also aims to determine the effectiveness of monthly injections of Sublocade® compared to daily oral Suboxone® SL therapy in the treatment of moderate to severe opioid use disorder after twenty-four weeks of treatment.

DETAILED DESCRIPTION:
While substance use disorders have been found to have relapse rates on part with other chronic illnesses such as hypertension and asthma long term abstinence remains elusive for many. Fortunately, the FDA has recently approved a long acting subcutaneous injectable formulation of buprenorphine. While this drug has proven effective in retaining patients in care and decreasing drug cravings as compared to placebo, this drug has not been tested in a real world clinic setting and no studies exist comparing it to the current formulations of buprenorphine. The objective of this study is to perform a randomized pilot study directly comparing sublingual buprenorphine/naloxone to long acting buprenorphine subdermal injection in a standard Office-Based Opioid Agonist Treatment (OBOT) clinic. The study team will compare patient retention, percentage of negative urinary drug screens, and withdrawal scores between the two groups. The findings will provide insight for US providers seeking more effective and efficient ways to treat Opioid use disorder (OUD) in the outpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who present to the WFBMC Medication-Assisted-Therapy (MAT) clinic seeking OBOT.

Exclusion Criteria:

* Those patients who have:
* history of cirrhosis, >= CKD stage 3
* congenital long QT syndrome
* those on antiarrhythmic medications
* liver enzymes more than 2 times the upper normal value at baseline assessment
* elevated bilirubin
* chronic pulmonary condition
* current unstable and untreated psychiatry comorbid disorder
* pregnant
* use of benzodiazepines/other CNS depressant medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of Weeks patients continued in treatment during trial period | 26 weeks
  Retention in weeks
Number of Participants that Dropout during the first 28 days of Treatment | first 28 days
  Number of participants that leave the study
Number of participants that complete of the treatment phase | 26 weeks
  Number of participants that complete the study
Number of participants who did not complete the trial in their assigned group | 26 weeks
  Total number of participants that changed arms
Percentage of negative urinary drug screens | 26 weeks
  percentage of participants that have a negative drug screen
Liver enzyme values - ALP, AST, ALT | 26 weeks
  Values of liver enzymes will be measured: Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST), and Alanine Aminotransferase (ALT). Values will be reported in IU/L
Liver enzyme values- Total Bilirubin | 26 weeks
  Values of liver enzymes will be measured: Total Bilirubin. Values will be reported in mg/dL
Clinical Opiate Withdrawal Scale (COWS) scores trends | 26 weeks
  Withdrawal symptoms scale- total score 0-48 with a lower score denoting no symptoms (better Outcomes) and higher score denoting more withdrawal symptoms
Subjective Opiate Withdrawal Scale (SOWS) score trends | 26 weeks
  Participant survey for how they are feeling during withdrawal period, score range from 0 to 64. Low score denotes no/less perceived symptoms (better outcomes) and higher score denotes high/ more personal perceived symptoms.
Number or patients still in medication assisted therapy (MAT) clinic 6 months after trial period ends. | 6 months
  Number of patients still in MAT clinics at 6 months
Number of participants death | 6 months
  Number of Participants deaths 6 months after initial participant consent is given.as measured by Vital Statistics database

CONTACTS AND LOCATIONS:
Overall Officials: Erin Barnes, MD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rudd RA, Aleshire N, Zibbell JE, Gladden RM. Increases in Drug and Opioid Overdose Deaths--United States, 2000-2014. MMWR Morb Mortal Wkly Rep. 2016 Jan 1;64(50-51):1378-82. doi: 10.15585/mmwr.mm6450a3. PMID 26720857
- [Background] Prevention CfDCa. Heroin Overdose Data. US Department of Health and Human Services. https://www.cdc.gov/drugoverdose/data/heroin.html. Published Jan 2017. Updated 2018-08-31T12:47:34Z. Accessed September 3 2018.
- [Background] Rudd RA, Seth P, David F, Scholl L. Increases in Drug and Opioid-Involved Overdose Deaths - United States, 2010-2015. MMWR Morb Mortal Wkly Rep. 2016 Dec 30;65(50-51):1445-1452. doi: 10.15585/mmwr.mm655051e1. PMID 28033313
- [Background] Fleischauer AT, Ruhl L, Rhea S, Barnes E. Hospitalizations for Endocarditis and Associated Health Care Costs Among Persons with Diagnosed Drug Dependence - North Carolina, 2010-2015. MMWR Morb Mortal Wkly Rep. 2017 Jun 9;66(22):569-573. doi: 10.15585/mmwr.mm6622a1. PMID 28594786
- [Background] Zibbell JE, Iqbal K, Patel RC, Suryaprasad A, Sanders KJ, Moore-Moravian L, Serrecchia J, Blankenship S, Ward JW, Holtzman D; Centers for Disease Control and Prevention (CDC). Increases in hepatitis C virus infection related to injection drug use among persons aged </=30 years - Kentucky, Tennessee, Virginia, and West Virginia, 2006-2012. MMWR Morb Mortal Wkly Rep. 2015 May 8;64(17):453-8. PMID 25950251
- [Background] Peters PJ, Pontones P, Hoover KW, Patel MR, Galang RR, Shields J, Blosser SJ, Spiller MW, Combs B, Switzer WM, Conrad C, Gentry J, Khudyakov Y, Waterhouse D, Owen SM, Chapman E, Roseberry JC, McCants V, Weidle PJ, Broz D, Samandari T, Mermin J, Walthall J, Brooks JT, Duwve JM; Indiana HIV Outbreak Investigation Team. HIV Infection Linked to Injection Use of Oxymorphone in Indiana, 2014-2015. N Engl J Med. 2016 Jul 21;375(3):229-39. doi: 10.1056/NEJMoa1515195. PMID 27468059
- [Background] Drug Enforcement Administration, Department of Justice.. Implementation of the Provision of the Comprehensive Addiction and Recovery Act of 2016 Relating to the Dispensing of Narcotic Drugs for Opioid Use Disorder. Final rule. Fed Regist. 2018 Jan 23;83(15):3071-5. PMID 29359892
- [Background] Public policy statement on Office-Based Opioid Agonist Treatment (OBOT). J Addict Dis. 2005;24(3):153-61. doi: 10.1300/J069v24n03_12. No abstract available. PMID 16186090
- [Background] Hser YI, Saxon AJ, Huang D, Hasson A, Thomas C, Hillhouse M, Jacobs P, Teruya C, McLaughlin P, Wiest K, Cohen A, Ling W. Treatment retention among patients randomized to buprenorphine/naloxone compared to methadone in a multi-site trial. Addiction. 2014 Jan;109(1):79-87. doi: 10.1111/add.12333. Epub 2013 Oct 9. PMID 23961726
- [Background] Kakko J, Svanborg KD, Kreek MJ, Heilig M. 1-year retention and social function after buprenorphine-assisted relapse prevention treatment for heroin dependence in Sweden: a randomised, placebo-controlled trial. Lancet. 2003 Feb 22;361(9358):662-8. doi: 10.1016/S0140-6736(03)12600-1. PMID 12606177
- [Background] Yokell MA, Zaller ND, Green TC, Rich JD. Buprenorphine and buprenorphine/naloxone diversion, misuse, and illicit use: an international review. Curr Drug Abuse Rev. 2011 Mar;4(1):28-41. doi: 10.2174/1874473711104010028. PMID 21466501
- [Background] Winchell C. Cross-Discipline Team Leader Review and Summary Basis for Approval. In: Administration FD, ed: Federal Drug Administration; 2017.
- [Background] (2017) USFDA. Press Announcements - FDA approves first once-monthly buprenorphine injection, a medication-assisted treatment option for opioid use disorder. 2018.
- [Background] Johnson RE, Chutuape MA, Strain EC, Walsh SL, Stitzer ML, Bigelow GE. A comparison of levomethadyl acetate, buprenorphine, and methadone for opioid dependence. N Engl J Med. 2000 Nov 2;343(18):1290-7. doi: 10.1056/NEJM200011023431802. PMID 11058673
- [Background] Surgeon General's Report: Facing Addiction in America. In: Services USDoHaH, ed. 200 Independence Avenue SW Washington DC 20201: U.S. Department of Health and Human Services; 2017.
- [Background] Park-Lee E, Lipari RN, Hedden SL, Kroutil LA, Porter JD. Receipt of Services for Substance Use and Mental Health Issues Among Adults: Results from the 2016 National Survey on Drug Use and Health. 2017 Sep. In: CBHSQ Data Review. Rockville (MD): Substance Abuse and Mental Health Services Administration (US); 2012-. Available from http://www.ncbi.nlm.nih.gov/books/NBK481724/ PMID 29431966
- [Background] McLellan AT, Lewis DC, O'Brien CP, Kleber HD. Drug dependence, a chronic medical illness: implications for treatment, insurance, and outcomes evaluation. JAMA. 2000 Oct 4;284(13):1689-95. doi: 10.1001/jama.284.13.1689. PMID 11015800
- [Background] Mattick RP, Breen C, Kimber J, Davoli M. Buprenorphine maintenance versus placebo or methadone maintenance for opioid dependence. Cochrane Database Syst Rev. 2014 Feb 6;2014(2):CD002207. doi: 10.1002/14651858.CD002207.pub4. PMID 24500948
- [Background] Jones CM, Campopiano M, Baldwin G, McCance-Katz E. National and State Treatment Need and Capacity for Opioid Agonist Medication-Assisted Treatment. Am J Public Health. 2015 Aug;105(8):e55-63. doi: 10.2105/AJPH.2015.302664. Epub 2015 Jun 11. PMID 26066931
- [Background] Rosenblatt RA, Andrilla CH, Catlin M, Larson EH. Geographic and specialty distribution of US physicians trained to treat opioid use disorder. Ann Fam Med. 2015 Jan-Feb;13(1):23-6. doi: 10.1370/afm.1735. PMID 25583888